CLINICAL TRIAL: NCT01887899
Title: Influence of Transcranial Direct-current Stimulation on Cortical Plasticity in Patients With Dementia of the Alzheimer Type
Brief Title: Influence of tDCS on Cortical Plasticity in Patients With Dementia of the Alzheimer Type
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Plasticity in Alzheimer's
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Dementia of Type Alzheimer
Keywords: cortical plasticity; transcranial direct current stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial direct current stimulation (Experimental)
  Interventions: Device: transcranial direct current stimulation
- sham stimulation (Placebo Comparator)
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation
  Arms: transcranial direct current stimulation
Device: sham stimulation
  Arms: sham stimulation

SUMMARY:
The aim of this study is to investigate whether the anodal transcranial direct current stimulation (tDCS) over the primary motor cortex (M1) in patients with dementia of the Alzheimer type (DAT) leads to an increase in cortical plasticity (change in motor evoked potentials (MEP) in mV).

ELIGIBILITY:
Inclusion Criteria:

* Right-handed according to the Oldfield Händigkeits inventory (lateralization index> 70) (1971)
* Cognitive impairment, which corresponds to a mild to moderate DAT
* No treatment with AChE inhibitors, or existing stable treatment with AChE inhibitors for over 3 months
* No motor impairments relevant to everyday life
* Age 50 to 80 years
* Existing Insurance certificate
* Existing informed consent

Exclusion criteria:

* Severe neurological / psychiatric or pre-existing internist conditions because additional cognitive deficits are expected
* Epilepsy, epileptic seizure in medical history
* Cognitive deficit (MMSE <20)
* Depressive episode (Beck Depression Inventory (BDI)> 12)
* intake of centrally active drugs <3 months, particularly acetylcholinesterase inhibitors
* Pregnancy
* Pacemaker (contraindication for MRI)
* Other metal parts in the body (contraindication for MRI)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the anodal transcranial direct current stimulation over the primary motor cortex (M1) in patients with dementia of Alzheimer type (DAT) | 1 week
  to investigate whether the anodal transcranial direct current stimulation over the primary motor cortex (M1) in patients with dementia of Alzheimer type (DAT) increases cortical plasticity (measured via motor evoked potentials) compared to a sham stimulation

SECONDARY OUTCOMES:
tDCS effects on central cholinergic activity in patients with DAT | 1 week
  to investigate whether the anodal transcranial direct current stimulation affect central cholinergic activity (measured via a TMS-protocol) in patients with dementia of Alzheimer type (DAT) compared to a sham stimulation
tDCS effects on learning | 1 week
  tDCS-induced changes in learning success (performance in a motor learning paradigm in patients with DAT after tDCS vs. sham stimulation)
MR elastography | 1 week
  Comparison of viscoelastic parameters in cerebral MR elastography in patients with DAT
genetic polymorphism, ApoE4 | once
  optional assessment of genetic Apo4 epsilon status for assessment of differences in cortical plasticity and elasticity between Apo4 epsilon positive and negative participants

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Neurologie, Charité Universitätsmedizin Berlin, Berlin, Germany